CLINICAL TRIAL: NCT02046031
Title: Preliminary Study of Pharmacokinetics of Ginkgolides Meglumine Injection.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z-YXPU-ZS-IV3
Record Dates: First submitted 2014-01-19; First posted 2014-01-27 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2013-12

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; safety; Pharmacokinetics; Ginkgolides Meglumine Injection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ginkgolides Meglumine Injection (Experimental): Intravenous drip slowly. A 1 (25 mg), will be taken slowly into the 0.9% sodium chloride injection diluted in 250 ml before use, then slow intravenous drip, once a day. The dripping speed must be strictly controlled. For the first time when using Ginkgolides Meglumine Injection, dripping speed should be controlled for 10 ~ 15 drops per minute. After 30 minutes treatment without discomfort, dripping speed can be appropriately increased, but no more than 30 drops per minute.
  Interventions: Drug: Ginkgolides Meglumine Injection

INTERVENTIONS:
Drug: Ginkgolides Meglumine Injection — 25 mg, ivdrip, once.

SUMMARY:
To explore the rule of absorption, distribution, metabolism and elimination after intravenous administration of Ginkgolides Meglumine Injection healthy subjects. The plasma drug profiles will be important to assess the potential clinical drug-drug interactions.

DETAILED DESCRIPTION:
Ginkgolides Meglumine Injection was jointly developed by China Pharmaceutical University and Jiangsu Kanion Pharmaceutical Co., Ltd. Its pharmacal ingredients are ginkgo lactones A , ginkgo lactone B, ginkgo lactone K, etc; Excipients for meglumine, citric acid, sodium chloride. It is used to treat stroke (mild-to-moderate cerebral infarction) in recovery phlegm and Syndrome of Intermingled Phlegm and Blood Stasis.

The aim of this study is to explore the rule of absorption, distribution, metabolism and elimination after intravenous administration of Ginkgolides Meglumine Injection healthy subjects. The plasma drug profiles will be important to assess the potential clinical drug-drug interactions.

Biological sample including blood and urine for PK is collected during the study. In the first stage, the biological sample of two subjects will be collected at different time points. In the second stage, the biological sample of another two subjects will be collected at the time points which are adjusted according to the results of the first stage.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-40, no more than 10 years apart.
* Both male and female.
* Subjects have standard weight( generally not less than 50 kg), and body mass index (BMI) within 19-25. Subjects weight (kg) should not differ too much.
* All physical examinations( including ECG, kidney function, liver function

  , blood routine, urine routines, etc) are normal.
* History of disease: no history of diseases in gastrointestinal tract, reproductive tract, urinary tract, heart, liver, kidney, lung, nervous system, metabolism, and no history of allergies and orthostatic hypotension.
* After being told all possible adverse reactions associated with the drug, subjects sign the informed consent and promise to complete all examinations.

Exclusion Criteria:

* Subjects who cannot communicate with medical staff, and subjects with cerebral insufficiency or psychological problem.
* Female subjects or partner of male subjects have plan to pregnant.
* Subjects have primary disease in significant organ.
* Subjects have history of drug dependence or psychosis in last 2 years.
* Subjects have blood loss or blood donation more than 200 mL 3 months prior to the baseline.
* Subjects who have taken part in other clinical trials 3 months prior to the baseline.
* Subjects who abuse alcohol or other drugs.
* Pregnancy or breast-feeding subjects.
* Subjects is found to have clinical significance of abnormal after checking information and physical examinations.
* Known allergies or serious side effects with no more than two kinds of food and drugs in the past.
* Subjects who have taken any drug during the previous 2 weeks.
* Subjects have unexplained infections.
* The subjects could not complete the study in the opinion of the Principal Investigator due to any reason.
* Positive HIV、HCV and HBsAg test results.
* A female subject whose pregnancy test is positive.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0, 4 days.
  Blood will be drawn from adult subjects pre-drug application and at 30min, 60min, 90min, 150min, 197min, 205min, 215min, 240min (4h), 300min(5h), 360min (6h), 480min (8h）， 720min (12h)，1440min(24h)，2160min(36h)， 2880min (48h)， 4320min (72h). Urine will be drawn from adult subjects pre-drug application and at 0-4, 4-6, 6-12, 12-24, 24-48, 48-72.
Time to maximum plasma concentration (Tmax) | 0, 4 days.
  Biological sample including blood, urine, faeces for PK will be collected at the same time point.
Area under the curve (AUC) | 0, 4 days.
  Biological sample including blood, urine, faeces for PK will be collected at the same time point.
Elimination half-life (t1/2) | 0, 4 days.
  Biological sample including blood, urine, faeces for PK will be collected at the same time point.
clearance (CL) | 0, 4 days.
  Biological sample including blood, urine, faeces for PK will be collected at the same time point.
Volume of distribution (Vd) | 0, 4 days.
  Biological sample including blood, urine, faeces for PK will be collected at the same time point.

SECONDARY OUTCOMES:
Safety assessments will be based on adverse event reports and the results of vital sign measurements, electrocardiogram, Electrocardiogram monitoring and clinical laboratory tests. | 0, 4days
  Adverse event reports will be assessed at 0, 4 days. Vital sign measurements will be assessed at pre-drug application and 30min, 60mi, 120min, 197min, 4h, 12h, 24h, 48h, 72h after application. Electrocardiogram will be assessed at 0, 4 days. Electrocardiogram monitoring will be assessed during medication period. Clinical laboratory tests will be assessed at 0, 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ou Ning, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital with Nanjing Medical University, Nanjing, Jiangsu, China